CLINICAL TRIAL: NCT07164079
Title: Effect of Dietary Supplementation of Rubus Sanctus (Wild Blackberry) Root Extract on Disease Prognosis in Graves' Disease: A Randomized Controlled Clinical Trial
Brief Title: Rubus Sanctus (Wild Blackberry) Root Extract as a Dietary Supplement for Graves' Disease
Acronym: RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Betul Uner (Other)
Responsible Party: Sponsor-Investigator, Betul Uner, Lecturer, MSc, Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-40160-152
Record Dates: First submitted 2025-08-25; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Graves Disease (Basedow's Disease)
Keywords: Rubus sanctus; Basedow disease; Toxic diffuse goiter; HEI
MeSH Terms: conditions — Graves Disease | interventions — Tea

STUDY DESIGN:
Intervention Model Description: Patients with newly diagnosed or recurrent Graves' disease will receive an 8-week intervention. Graves' disease patients assigned to the control group will be asked to consume black tea (Camellia sinensis) with their breakfast for 8 weeks. The black tea will be prepared as 5 g doses and steeped in 200 ml of water at 80 °C for 5 minutes. The intervention group will be given Rubus Sanctus root extract, which they will consume with breakfast for 8 weeks. The tea will be packaged as 5 g Rubus Sanctus root and steeped in 200 ml of water at 80 °C for 5 minutes. Participants in the intervention and control groups will receive black tea and Rubus Sanctus root tea, along with the necessary equipment (a 200 ml beaker and a thermometer).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blackberry root group (Experimental): Patients in the intervention group will receive a Rubus Sanctus root extract, which they will consume with breakfast for 8 weeks.
  Interventions: Dietary Supplement: blackberry root
- Black Tea group (Placebo Comparator): Patients with Graves' disease assigned to the control group will be asked to consume black tea (Camellia sinensis) with their breakfast for 8 weeks.
  Interventions: Dietary Supplement: black tea

INTERVENTIONS:
Dietary Supplement: blackberry root — Patients in the intervention group will receive a Rubus Sanctus root extract, which they will consume with breakfast for 8 weeks. The tea will be packaged as 5 grams of Rubus Sanctus root and steeped in 200 ml of water at 80°C for 5 minutes. Participants in the intervention group will receive the Rubus Sanctus root tea along with the necessary equipment (a 200 ml beaker and thermometer). Measurements of TSH, T4, T3, anti-TPO, anti-TG, TSH receptor antibodies, liver function tests, thyroid parenchymal echogenicity, and thyroid volume will be taken at the Endocrinology and Metabolic Diseases Clinic of Muğla Training and Research Hospital before and after the study.
  Arms: Blackberry root group
Dietary Supplement: black tea — Patients with Graves' disease assigned to the control group will be asked to consume black tea (Camellia sinensis) with their breakfast for 8 weeks. Black tea is a product consumed almost daily in Turkish society. Black tea will be prepared in 5-g doses and steeped in 200 ml of water at 80°C for 5 minutes. Participants in the control group will be provided with black tea bags along with the necessary equipment (a 200 ml beaker and thermometer). TSH, T4, T3, anti-TPO, anti-TG, TSH receptor antibody, liver function tests, thyroid parenchymal echogenicity, and thyroid volume will be obtained before and after the study at the Endocrinology and Metabolic Diseases Clinic of Muğla Training and Research Hospital.
  Arms: Black Tea group

SUMMARY:
The aim of this single-blind, randomized, experimental study was to investigate the effect of Rubus sanctus root extract, which has antioxidant properties, added to the routine diet of patients with Graves' disease on the prognosis of the disease.

The study sample included patients who presented to the Endocrinology and Metabolic Diseases Outpatient Clinic of Muğla Sıtkı Koçman University Training and Research Hospital and were diagnosed with Graves' disease or developed a relapse after necessary examinations. Cohen's standardized effect size was used. Accordingly, the required sample size for the study was determined to be 42, using an alpha value of 0.05, an effect size of 0.80, and a theoretical power of 80%. The study planned to include a minimum of 42 participants: 21 intervention participants and 21 controls.

Patients assigned to the control group were asked to continue their routine diet, adhere to any necessary pharmacological treatments, and consume a placebo tea for the planned 8-week intervention period. Routine monthly examinations will be collected, and anthropometric measurements will be repeated at the end of 8 weeks.

Patients assigned to the experimental group will be asked to continue their routine diet for 8 weeks, comply with any required pharmacological treatments, and consume Rubus sanctus root extract, produced by aqueous extraction and lyophilization, with active ingredient (phenolic compound) determined by LC-MS-MS, and prepared as a tea in 5-g packets. Anthropometric measurements will be repeated at the end of 8 weeks.

H0: Rubus sanctus root extract supplemented to the diet has no effect on Graves' disease.

H1: Rubus sanctus root extract supplemented to the diet has an effect on Graves' disease.

DETAILED DESCRIPTION:
Humanity has fought many battles for survival. One of the most important of these battles is the fight against disease. The imbalance between free radicals and antioxidants in the body leads to oxidative stress, which in turn contributes to a range of diseases, including autoimmune diseases. To avoid diseases that may arise from oxidative stress, it is recommended that individuals ensure they consume adequate amounts of antioxidants in their routine diet, avoid harmful habits that increase oxidant production, such as smoking and alcohol, exercise regularly, and get adequate sleep.

Since ancient times, various parts of plants have been used to treat illnesses. The blackberry plant, with its fruit, leaves, stem, and root, is considered one of these plant products. The blackberry plant belongs to the Rubus genus of the Rosaceae family. Rubus sanctus is the most common species in the Muğla region. Wild blackberries are strong, thorny shrubs that grow primarily in forests, vacant lots, and along roadsides. The fruit is usually black and edible. It is reported in the literature that extracts of the aboveground parts of the blackberry plant are used to heal infected insect bites and skin wounds, teas obtained from the plant roots are used in the autoimmune disease rheumatoid arthritis and to relieve pain, and extracts obtained from the leaves and roots are used in diarrhea due to their antimicrobial effects.

The beneficial health effects of blackberry root extract are attributed to its polyphenol content. The polyphenols found in blackberry root extract include the phenolic acids gallic acid, the flavonoids quercetin, apigenin, and catechins, the tannins ellagic acid, the terpenes triterpenes, including betulinic acid, which has anti-carcinogenic effects, and α-tocopherol.

Mice studies have determined that different doses of blackberry root extract have anti-inflammatory properties, promote wound healing and skin symptoms, and exhibit neuropharmacological effects. Another study reported that blackberry root extract exhibits antibacterial activity against Staphylococcus aureus. An in vitro study demonstrated that blackberry root (Rubus sanctus) extract possesses potential anticancer, antioxidant, anti-lipase, and α-amylase inhibitory activity. The study concluded that blackberry root extract may be a promising resource for applications in the functional food, nutraceutical, and pharmaceutical industries.

Autoimmune thyroid diseases are defined as a group of diseases in which the immune system targets and attacks the thyroid gland. These diseases include Hashimoto's thyroiditis and Graves' disease, and have two extreme clinical presentations. Both conditions are characterized by thyroid dysfunction, but they differ in their pathogenesis and clinical symptoms. There is evidence in the literature that the COVID-19 pandemic has led to an increase in autoimmune thyroid diseases. The global prevalence of autoimmune thyroid diseases varies depending on geographic, ethnic, and environmental factors. However, these diseases are considered a significant health problem worldwide and are, on average, 5-7 times more common in women. The prevalence of Graves' disease ranges from 0.5% to 1.0%.

Graves' disease is a hyperthyroidism condition characterized by an overactive thyroid gland and excessive production of thyroid hormone. In this disease, thyroid-stimulating hormone (TSH) autoantibodies (TSH) are produced against the TSH receptor. These antibodies activate the thyroid-stimulating hormone (TSH) receptor, causing the thyroid gland to continuously and uncontrollably produce thyroid hormones. Clinical symptoms of Graves' disease include ophthalmopathy, palpitations, hand tremors, excessive sweating, weight loss, irritability, and sleep problems. Diagnosis is based on clinical findings, hormone levels measured through blood tests, and the presence of autoantibodies. Treatment for Graves' disease may include antithyroid medications, radioactive iodine therapy, or surgery.

Providing nutritional therapy in addition to medical treatment is crucial for individuals with Graves' disease. The importance of antioxidant and anti-inflammatory nutrition, which can help reduce the inflammation underlying autoimmune diseases, is well known. In this regard, a randomized controlled trial was conducted in which broccoli sprout extract, high in sulforaphane, was administered to patients with Graves' disease for 12 weeks. The study reported that the broccoli sprout extract beverage had no detrimental effects on thyroid function tests or thyroid autoimmunity measurements and provided protection against pathologies associated with oxidative stress and inflammation. Yingliu is a mixture of the antioxidant plants found in Chinese medicine, consisting of the following: Radix astragali Leguminosae, Radix scrophulariae Scrophulariaceae, Radix ophiopogonis, Ophiopogon japonicus, Rhizoma anemarrhenae Liliaceae, Fructus forsythiae Oleaceae, Spica prunellae Labiatae, Concha ostreae Ostreidae, and Bulbus fritillariae thunbergii Liliaceae. Yingliu is widely used in the treatment of Graves' disease and has yielded positive results.

The increasing prevalence of autoimmune thyroid diseases necessitates the search for new solutions. It is recognized that autoimmune thyroid diseases are a global health problem and that comprehensive health strategies must be developed for the management of these conditions. Early diagnosis and appropriate treatment, especially in at-risk groups, are critical to preventing disease-related complications. Evidence in the literature indicates that different parts of plants have positive effects on diseases, and the roots of plants, in particular, have been traditionally used throughout history. Therefore, the aim of our study was to investigate the effects of Rubus sanctus root extract, a wild blackberry species with antioxidant properties, added to the routine diet of Graves' patients on serum thyroid hormone and disease-related symptoms.

This experimental randomized controlled study, planned as a controlled trial, initiated face-to-face data collection after receiving ethics committee approval. Four- and six-way block randomization was used to ensure randomization. Patients were randomized to experimental and control groups at a 1:1 ratio.

The Cohen-standardized effect size was used to calculate the study's sample size. Accordingly, the required sample size for the study was determined to be 42, using an alpha value of 0.05, an effect size of 0.80, and a theoretical power of 80%. The study planned to include 42 individuals, 21 as intervention and 21 as controls. The study sample included patients aged 18-65 who presented to the Endocrinology and Metabolic Diseases Outpatient Clinic of Muğla Sıtkı Koçman University Training and Research Hospital, were diagnosed with Graves' disease or developed relapse after the necessary tests, and scored at least 80 on the Healthy Eating Index (HEI). The 24-hour individual food consumption method will be used to assess nutritional status. The average energy and nutrient values of consumed foods will be calculated using the "Computer Assisted Nutrition Program, Nutrition Information System (BEBIS)" (BEBIS 4.). The HEI-2015 index includes 12 healthy nutrition components: total fruit (5 points); whole fruit (5 points); total vegetables (5 points); dark green and orange vegetables and legumes (5 points); total grains (5 points); whole grains (5 points); milk (10 points); meat products and legumes (10 points); fats (10 points); saturated fat (10 points); sodium (10 points); and calories from solid fats, alcoholic beverages (beer, wine, and spirits), and added sugars (20 points), and has a total score of 100. An individual with an HEI score of 80 and above is classified as "good" in terms of diet quality.

Participants who agree to participate in the study and meet the inclusion criteria will have their monthly tests (TSH, T4, T3, anti-TPO, anti-TG, TSH receptor antibody, and liver function tests) routinely requested by the Endocrinology and Metabolic Diseases Polyclinic of Muğla Sıtkı Koçman University Training and Research Hospital. These tests will be collected in person after receiving approval from the ethics committee. Thyroid parenchymal echogenicity and thyroid volume will be assessed before and after the study using a thyroid ultrasound in the Endocrinology and Metabolic Diseases Clinic. These routine tests will monitor the effects of the intervention on disease serum hormone levels and symptoms. Patient anthropometric measurements will be taken by researchers in the Research Laboratory of the Department of Nutrition and Dietetics, Faculty of Health Sciences, Muğla Sıtkı Koçman University. Patient body composition will be determined using a Tanita SC 330 BIA device. Circumference measurements will be measured in three areas (neck, waist, and hips) using a 0.5 cm wide, non-stretchable tape measure. Height will be measured in the Frankfort plane (head upright, eyes looking forward, body upright, arms relaxed at sides) with a portable height meter capable of measuring between 14 and 200 cm with an accuracy of 0.1 cm.

Patients assigned to the control group will be asked to continue their routine diet, comply with any necessary pharmacological treatments, and consume black tea (Camellia sinensis), a staple in Turkish culture, for the planned 8-week intervention period. Routine monthly tests will be collected, and anthropometric measurements will be repeated at the end of the 8 weeks. Patients assigned to the experimental group will continue their routine diet for 8 weeks, adhere to any necessary pharmacological treatments, and take a daily supplement of 5 g of Rubus sanctus root extract in tea form, which was produced by aqueous extraction and lyophilization, and whose active ingredient (phenolic compound) content was determined by LC-MS-MS. The Rubus sanctus root extract in tea form will be provided to the participants by the researchers. Animal studies have shown no toxic effects of Rubus sanctus root extract. Patients will be interviewed weekly in person or by phone to obtain feedback on any potential product discontinuation, to determine toxicity, and to discontinue the study. Anthropometric measurements will be repeated at the end of the 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a new diagnosis of Graves' disease or those with a relapse of Graves' disease
* Patients aged 18-65
* A score of 80 or higher on the Health Eating Index (HEI)

Exclusion Criteria:

* Having received treatment for the disease within the last 6 months
* Having another chronic and/or autoimmune disease
* Being pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Effect of Rubus sanctus root on thyroid hormones | 8-week intervention
  It will be determined whether the use of Rubus sanctus in Graves' patients causes changes in the blood parameters of the thyroid hormones TSH, T4, and T3 associated with the disease.
Effect of Rubus sanctus use on disease-related autoimmune markers | 8-week intervention
  It will be determined whether the use of Rubus sanctus in Graves' disease patients causes changes in blood parameters such as anti-TPO, anti-TG, and TSH receptor antibodies, which are autoimmune markers associated with the disease.
Determination of anatomical and structural changes in the thyroid gland due to the use of Rubus sanctus | 8-week intervention
  The effect of Rubus sanctus use on thyroid parenchymal echogenicity and thyroid volume in Graves' disease will be determined by thyroid ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Betül Üner Yılmaz, Lecturer, Principal Investigator — https://www.mu.edu.tr/tr/personel/betuluner
Locations (1):
- Muğla Sıtkı Koçman University/Muğla Training and Research Hospital Endocrine and Metabolic Diseases Polyclinic, Muğla, Mentese, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data obtained as a result of the study will be presented in a report form.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: December 2024 - December 2026

REFERENCES:
- [Background] Yang H, Bi X, Tang H, Zeng J, Cong Y, Wu T, Chen Q. Clinical efficacy of Yingliu treatment for Graves disease. Int J Clin Exp Med. 2015 Apr 15;8(4):6145-53. eCollection 2015. PMID 26131218
- [Background] Jaradat N, Dwikat M, Amer J, Hawash M, Hussein F, Qneibi M, Issa L, Asab JA, Hallak H, Arar DN, Masri HZ, Obeid K, Sharabati M, Kittaneh R. Anticancer, Free Radicals, and Digestive Enzyme Inhibitory Activities of Rubus sanctus Schreb Root Four Solvent Fractions. Evid Based Complement Alternat Med. 2021 Jun 16;2021:6690646. doi: 10.1155/2021/6690646. eCollection 2021. PMID 34221089